CLINICAL TRIAL: NCT04905147
Title: Randomized Controlled Trials of Efficacy of Mosapride on Recovery of Intestinal Motility After Elective Colorectal Cancer Surgery
Brief Title: Efficacy of Mosapride on Recovery of Intestinal Motility After Elective Colorectal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COA.MURA2021/328
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Bowel Ileus
Keywords: Postoperative ileus; Colorectal Cancer Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Ileus | interventions — mosapride

STUDY DESIGN:
Intervention Model Description: The mosapride group received 15 mg of mosapride by mouth or feeding via NG with 50 ml of water three times a day, starting on the morning of postoperative day 1, until hospital discharge or for a maximum of 10 postoperative days if the patient remained hospitalized.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The mosapride group (Active Comparator): The mosapride group received 15 mg of mosapride by mouth or feeding via NG with 50 ml of water three times a day, starting on the morning of postoperative day 1, until hospital discharge or for a maximum of 10 postoperative days if the patient remained hospitalized.
  Interventions: Drug: Mosapride
- The control group (Placebo Comparator): The control group received 15 mg of placebo drug with 50 ml of water three times a day, starting on the morning of postoperative day 1, until hospital discharge or for a maximum of 10 postoperative days if the patient remained hospitalized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mosapride — Mosapride citrate is prokinetic drug that selectively activates 5-HT4receptors. Mosapride stimulates serotonin receptor in the digestive tract and increases acetylcholine release to promote upper digestive tract (stomach and duodenum) and lower digestive tract (colon) motility and gastric emptying without cardiac side effects
  Other Names: The mosapride group
  Arms: The mosapride group
Drug: Placebo — Placebo drug 15 mg
  Other Names: The placebo group
  Arms: The control group

SUMMARY:
Postoperative ileus (POI) is one of the most common causes of prolonged hospital stays after abdominal surgery. The pathophysiology of POI is multifactorial and complex.It is known to be associated with sympathetic neural reflexes,local and systemic inflammatory mediators,and changes invarious neural and hormonal transmitters.Sympathetic (adrenergic) hyperactivity results in reduction of propulsive motility,and an increase in sphinctertone.Parasympathetic (cholinergic) hypoactivity results in adecrease in gastrointestinalmotility. Various agents called prokinetic drugs,including erythromycin, metoclopramide, cholinergic agents have been assessed in an effort to improved gastrointestinal motility. Mosapridecitrate is another prokinetic drug that selectively activates 5-HT4 receptors. Mosapride stimulates serotonin receptor in the digestive tract and increases acetylcholine release to promote upper digestive tract (stomach and duodenum) and lower digestive tract (colon) motility and gastric emptying without cardiac side effects. We therefore investigate the effect of mosapride on postoperative gastrointestinal motility after open and laparoscopic colectomy in a prospective randomized, controlled study in patients under going colectomy.

DETAILED DESCRIPTION:
This prospective blinded (participants,researchers,investigators) randomizedcontrolledtrial (RCT) is aimed to study the efficacy of the prokinetic agents, specifically, Mosapride on gastrointestinal recovery in patients under going colorectal cancer surgery. The patients are divided into two groups and each group will receive oral Mosapride and placebo,respectively. The primary outcome is to study the efficacy of Mosapride compared with placebo on gastrointestinal recovery in patients undergoing elective colorectal cancer surgery.

The participants were randomly assigned to receive mosapride (22patients) or to serve as placebo (22patients). Patients first were randomly assigned to one of the two groups. The mosapride group received 15 mg of mosapride by mouth or feeding via NG with 50 ml of water three times a day, starting on the morning of postoperative day 1, until hospital discharge or for a maximum of 10 postoperative days if the patient remained hospitalized. The control group received15 mg of placebo drug with 50ml of water on the same schedule.

Oral feeding was allowed when the first bowel sound and the first passage of flatus was came. A clear liquid diet is the first postoperative meal. If patient well tolerated, next step diet was applied (full liquid diet, soft diet, regular diet). Patients were discharged when the following criteria were fulfilled: 1) regular diet was tolerated without discomfort; 2) bowel movements had returned; and 3) body temperature was normal, with no major complications present.

The duration on first time bowel movement or first passage of flatus, postoperative hospital stay and adverse effects will be evaluated. The This trial was designed to have 90 percent power to detect a 20 percent decrease in median postoperative time to the first of bowel movement at a significance level of 5 percent. The necessary patient accrual to detect this difference was determined to be 20 patients per group and 10 % drop off was calculated so the totally patient was 22 patients per groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing elective colorectal cancer surgery at Ramathibodi hospital both open and laparoscopic surgery.
* Both male and female who age between 15 to 70 years old.
* Physical status American Society of Anesthesiologists (ASA) classification1-2-3.

Exclusion Criteria:

* Metastatic disease.
* Patients who reject to participate or withdrawal from the research.
* History of Mosapride allergy.
* Pregnancy.
* Emergency colorectal cancer surgery.
* Intestinal perforation or obstruction.
* Patients who have cardiac problem (Side effects of Mosapride may include arrhythmia or QTprolong).
* Physical status American Society of Anesthesiologists (ASA) classification 4-5.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative time to the first passage of flatus. | 24 hours
  Postoperative time to the first passage of flatus or the first bowel movement, as evaluated by one of the investigators (surgical resident) who was blinded as to whether the patient had received mosapride.
Postoperative time to the first passage of flatus. | 48 hours
  Postoperative time to the first passage of flatus or the first bowel movement, as evaluated by one of the investigators (surgical resident) who was blinded as to whether the patient had received mosapride.
Postoperative time to the first passage of flatus. | 72 hours
  Postoperative time to the first passage of flatus or the first bowel movement, as evaluated by one of the investigators (surgical resident) who was blinded as to whether the patient had received mosapride.

SECONDARY OUTCOMES:
Length of postoperative hospital stay | 30 day
  Length of postoperative hospital stay, and occurrence of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi hospital, Mahidol University.; Tharin Thampongsa, MD, Study Chair — Ramathibodi hospital, Mahidol University.; Bensita Saengsawang, MD, Principal Investigator — Ramathibodi hospital, Mahidol University.; Jakrapan Jirasiritham, MD, Study Director — Ramathibodi hospital, Mahidol University.
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thampongsa T, Saengsawang B, Supsamutchai C, Wilasrusmee C, Jirasiritham J, Punmeechao P, Palitnonkiat V, Poprom N, Choikrua P, Singhathas P. The efficacy of mosapride on recovery of intestinal motility after elective colorectal cancer surgery: a randomized controlled trial. Ann Coloproctol. 2025 Jun;41(3):232-238. doi: 10.3393/ac.2024.00892.0127. Epub 2025 Jun 25. PMID 40598989